CLINICAL TRIAL: NCT07072390
Title: Clinical Competence Measurement Tool in Physiotherapy (FKYÖA): Turkish Adaptation, Validity, and Reliability
Brief Title: Turkish Validation of Clinical Competence Tool in Physio
Acronym: CCMTP
Status: Completed | Type: Observational
Sponsor: University of Yalova (Other)
Responsible Party: Sponsor
Other Study IDs: CCMTP
Record Dates: First submitted 2025-07-05; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Reliability
Keywords: Clinical competence; Educational measurement; Professional practice; Physiotherapy and Rehabilitation; Students
MeSH Terms: interventions — Clinical Competence; Physical Therapy Modalities

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Physiotherapy Students Group: This is a non-interventional, cross-sectional observational study aimed at evaluating the psychometric properties of a clinical competence assessment tool among physiotherapy students.
  Interventions: Other: Measurement Tool for Clinical Competencies in Physiotherapy (MTCCP)

INTERVENTIONS:
Other: Measurement Tool for Clinical Competencies in Physiotherapy (MTCCP) — A culturally adapted Turkish version of the Measurement Tool for Clinical Competencies in Physiotherapy (MTCCP), used to evaluate clinical skills in final-year physiotherapy students.

SUMMARY:
In this study, the adaptation, validity and reliability of the Clinical Competence Measurement Tool in Physiotherapy (FKYÖA) in Turkish were examined. A total of 105 (female: 76, male: 29) senior students of the Department of Physiotherapy and Rehabilitation (FTR) aged between 21-25 with a mean age of 23.1 years were included in the study. Demographic information of the students participating in the study was recorded. In the process of translating the scale into Turkish, after the translation into Turkish, translation back into English and cultural adaptation process was completed, the suitability of each item in terms of comprehensibility, equivalence, suitability and representation of the content was evaluated with the expert opinions received from 10 faculty members working in the FTR departments of the relevant universities in order to examine the content validity (CGI: 1.0). Within the scope of the validity analysis of the scale, language, structure and scope validity were examined. Confirmatory Factor Analysis (CFA) was applied for construct validity. Within the scope of the reliability analysis of the scale, the test was applied 2 times with an interval of 10 days under similar conditions to 20 students who were randomly determined for the reliability of the test-retest and to evaluate the internal consistency. Cronbach's alpha coefficient was calculated.

ELIGIBILITY:
Inclusion Criteria:Final-year students enrolled in the Department of Physiotherapy and Rehabilitation at Karabük University or Yalova University

Aged between 21 and 25 years

Voluntary participation with signed informed consent

Able to read and understand Turkish fluently

Exclusion Criteria:

Students not in their final year of physiotherapy education

Individuals who did not provide informed consent

Incomplete or missing responses on the data collection forms

Inability to complete the scale due to cognitive or communication difficulties

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consisted of final-year undergraduate students enrolled in the Physiotherapy and Rehabilitation Departments at Karabük University and Yalova University. A total of 105 students (76 female and 29 male), aged between 21 and 25 years (mean age 23.1), voluntarily participated in the study. All participants were native Turkish speakers and met the inclusion criteria for assessment of clinical competence using the Turkish version of the MTCCP scale.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Construct Validity of the Turkish Version of the MTCCP (Measurement Tool for Clinical Competencies in Physiotherapy) | 1 month
  Structural validity assessed via Confirmatory Factor Analysis (CFA)
Internal Consistency Reliability of the MTCCP (Measurement Tool for Clinical Competencies in Physiotherapy) | 1 month
  Reliability evaluated using Cronbach's alpha coefficient across subscales.

CONTACTS AND LOCATIONS:
Locations (3):
- Turkey (Türkiye) (3):
  - Facility Name: Karabük University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Karabük, Karabük Province
  - asuman SALTAN, Yalova, Yalova
  - Yalova University, Yalova, Yalova

IPD SHARING:
Plan to Share IPD: No